CLINICAL TRIAL: NCT06963008
Title: A Prospective, Single-center, Open-label Clinical Study to Evaluate the Safety and Efficacy of Inhaled BMD003(CFTR mRNA) in Chinese Adult Patients With Cystic Fibrosis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xinlun Tian, Chief physician, professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMD003-001
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis (CF); Gene Therapy
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- inhaled BMD003(CFTR mRNA) (Experimental)
  Interventions: Drug: inhaled BMD003(CFTR mRNA)

INTERVENTIONS:
Drug: inhaled BMD003(CFTR mRNA) — BMD003 is the world's first freeze-dried CFTR Mrna product (stored at 2-8 ℃), which is reconstituted with injection water before use, nebulized through a vibrating sieve atomizer, and inhaled into the lungs through the mouth and nose.

SUMMARY:
The study adopts a prospective, single-center, open-label clinical study to evaluate the safety and efficacy of inhaled BMD003(CFTR mRNA) in Chinese adult patients with cystic fibrosis This study is a single dose escalation study of BMD003 nebulized inhalation in CF patients.

The study is divided into four cohorts, they are 2mg, 4mg, 8mg, and 16mg dose groups. The first dose group (2mg) is planned to enroll one patient. During the study, if there are ≥ 2 grade treatment-related adverse events (TRAEs) related to the investigational product that occur during the study period, 2 patients will be added at the current dose level. Each of the remaining groups will include 2-3 subjects, regardless of gender. Based on the safety data review of subjects in the previous dose group 4 weeks after administration, subjects in the next dose group will be allowed to receive the next higher dose, while patients in the previous dose group will complete the study.

The study includes three stages: screening period (2 weeks), administration period (1 day), and follow-up period (approximately 13 months). After passing the screening of the subjects, D1 was admitted to the hospital, D1 received a single nebulized inhalation investigational product (BMD003), and D2 completed safety observation before being discharged.

During the study, PK sample collection and safety assessment will be conducted at the corresponding visit points. After the treatment is completed, each patient will be followed up according to the schedule specified in the protocol.This study will conduct multiple dosing studies after the end of a single dose escalation. Multiple dosing doses, dosing intervals, etc. will be revised based on preclinical data and single dose data, and will be implemented after ethical approval.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be included in this study:

1. Gender not limited, 18 years old and above (including threshold values);
2. The subjects themselves agree to participate in the study and sign an informed consent form
3. Diagnosed with cystic fibrosis (CF);
4. According to the investigators' assessment, the subject's cystic fibrosis disease is clinically stable;
5. During screening, the subject's body mass index (BMI) is ≥ 17.5 kg/m ² and their weight is ≥ 40 kg;
6. Forced Expiratory Volume in 1 second (FEV1) is expected to be ≥ 40% of the normal value;
7. Resting oxygen saturation (SpO2) ≥ 92%;
8. Quit smoking for at least 2 years;
9. The subjects are willing and able to comply with the scheduled visits, treatments, laboratory tests, contraception requirements, and other study procedures.

Exclusion Criteria:

Individuals who meet any of the following criteria are not eligible for inclusion in this study:

1. Acute respiratory infection, acute exacerbation of lung disease, clinically significant hemoptysis (>30 mL, or as determined by the investigator), or changes in respiratory medications (including antibiotics, oral steroids, etc.) used to treat CF occurred within 4 weeks prior to the first administration;
2. Infected with highly virulent bacteria associated with accelerated decline in lung function and/or shortened survival time (e.g. Burkholderia cepacia, Mycobacterium abscesses). For subjects with a positive culture history, they can be considered uninfected according to the following guidelines:

   All culture results obtained in the past 12 months have been negative. Subject should have undergone at least 2 cultures within the past 12 months, with a minimum interval of 3 months between each culture, and at least one culture should have been conducted within 6 months prior to screening in this study.
3. During screening, the 12 lead electrocardiogram showed prolonged QTcF interval (>450 ms for males and>460 ms for females) and clinically significant abnormalities in other indicators of the 12 lead electrocardiogram.
4. During screening, total bilirubin exceeded the upper limit of normal, ALT and AST exceeded three times the upper limit of normal, and blood creatinine (CRE) was ≥ 1.5 times the upper limit of normal.
5. History of physical organ or blood transplantation or registered waiting for transplantation;
6. During screening, positive for human immunodeficiency virus antibodies (HIV Ab) and positive for Treponema pallidum specific antibodies (TPPA);
7. Participated in inhalation drug or device studies within 30 days prior to the initial screening visit (a 30 day window period applies to inhalation drugs with elimination half-life<6 days. If the elimination half-life of inhalation drugs is ≥ 6 days, the window period should be extended to at least 5 half lives after the last administration);
8. Pregnant (positive blood pregnancy test result) or lactating women;
9. Having a history of drug allergies or other allergies, which investigators consider to be contraindications for participation in the study;
10. History of drug allergies or other allergies, and investigators believe it contraindications for participation in the study;
11. Investigators believe that any medical indicators (including other laboratory test indicators with clinical significance) or other conditions that may affect clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2026-05-10 (Estimated); Study Completion 2027-05-10 (Estimated)

PRIMARY OUTCOMES:
Observe adverse events (AE) and serious adverse events (SAE) | From enrollment to the end of treatment at 13 months

SECONDARY OUTCOMES:
Expected percentage of forced expiratory volume in one second (ppFEV1) change from baseline | From enrollment to the end of treatment at 13 months
Changes in the revised cystic fibrosis questionnaire (CFQ-R score) compared to baseline | From enrollment to the end of treatment at 13 months

IPD SHARING:
Plan to Share IPD: No